CLINICAL TRIAL: NCT00562835
Title: Randomized, Placebo-Controlled, Double-Blind Clinical Trial to Evaluate the Safety and Efficacy of Low-Dose Glucocorticoid Infusion in Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Steroids in Patients With Early ARDS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Prot.cm.P662(A.1552)/C.E./2007
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Acute Lung Injury; ARDS, Human
Keywords: ARDS; Adult; Methylprednisolone
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Methylprednisolone; Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone
- 2 (Placebo Comparator)
  Interventions: Other: Normal saline intravenously and vitamin B1 per os

INTERVENTIONS:
Drug: Methylprednisolone — Drug: Methylprednisolone Day 0 Loading dose 1 mg/kg IV bolus (30 min) followed by continuous infusion; Days 0 to 14*† ‡ 1 mg/kg/day mixed in 240cc Normal saline (NS) and infused at 10 cc/hr; Days 15 to 21*‡ 0.5 mg/kg/day mixed in 240cc NS and infused at 10 cc/hr; Days 22 to 25*‡ 0.25 mg/kg/day; Days 26 to 28*‡ 0.125 mg/kg/day
  *Five days after the patient is able to ingest medications, methylprednisolone is given per os in one single daily equivalent dose.
  †If between days 1 to 14 the patient is extubated, he is advanced to day 15 of drug therapy and tapered according to schedule.
  ‡ When leaving ICU, if the patient is still not tolerating p.o. intake for at least five days, he should receive the specified dosage as IV push every 6 hours until tolerating oral ingestion
  Arms: 1
Other: Normal saline intravenously and vitamin B1 per os — Patients in this group will receive sterile normal saline in an amount that would equal the total diluted dose of study drug (ie. if initial loading dose equals a total of 25 cc [prednisolone + diluting fluid], then the patient will receive 25 cc of sterile normal saline). Tapering doses will be equivalent to that of the study arm. Five days after the patient is able to ingest medications, placebo is administered per os in one single daily equivalent dose. The placebo will be a Vitamin B1 (thiamine) 50-mg tablet. We will now designate each placebo tab as a 16-mg equivalent to each tablet of active drug. These tablets are scored and half tabs can be given if needed. Therefore if a patient is receiving 40 mg of study drug: 40/16 = 2.5 tabs x 50 mg = 125 mg actual dose of thiamine.
  Other Names: Thiamine
  Arms: 2

SUMMARY:
Scientific background. Dysregulated systemic inflammation is a key pathogenetic mechanism for morbidity and mortality in ALI/ARDS, and is associated with tissue insensitivity and/or resistance to inappropriately elevated endogenous glucocorticoids. In one study, prolonged methylprednisolone treatment of ARDS patients resulted in rapid and sustained reduction in circulating and pulmonary levels of pro-inflammatory cytokines, chemokines, and procollagen.

Preliminary work. Five randomized trials (N = 518) investigating prolonged glucocorticoid treatment in acute lung injury/ARDS reported a significant physiological improvement and a sizable reduction in duration of mechanical ventilation and ICU length of stay. Insufficient data is available on the effects of low dose prolonged methylprednisolone treatment initiated in early ALI/ARDS on mortality.

Hypothesis. We hypothesized that the anti-inflammatory activity associated with prolonged methylprednisolone administration improves pulmonary and extra-pulmonary organ dysfunction in early ALI/ARDS and reduces mortality.

Objective. To investigate the effects of prolonged low-dose methylprednisolone infusion on mortality and morbidity in early ALI/ARDS.

Study design. Multicenter, prospective randomized, placebo-controlled, double-blind clinical trial.

Entry criteria. Patients with ALI/ARDS of less than 72 hours duration.

Stratification. Patients are prospectively stratified prior to randomization as (1) intubated versus NPPV treated, and (2) ARDS versus severe ARDS. The purpose of stratification is to distribute equally in both arms intubated versus NPPV treated, and ARDS versus severe ARDS.

End-points. The primary end-point of trial is 28 days all cause mortality; the secondary end-points are (a) ventilator-free days at 28 days following study entry, (b) organ failure-free days at 28 days following study entry, and (c) duration of ICU stay.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND. Acute respiratory distress syndrome (ARDS) is a life-threatening form of acute hypoxemic respiratory failure that develops rapidly (12-48 hours), in the setting of an acute severe illness complicated by systemic inflammation.

Overall mortality in ARDS is 35-60%, with most nonsurvivors dying within two weeks of disease development. While a regulated inflammatory response is critical to survival, a major predictor of poor outcome in ARDS patients is persistence of pulmonary and systemic inflammation after one week of lung injury. Innate or treatment-induced downregulation of systemic inflammation is important to the resolution of ARDS.Failure to downregulate the production of inflammatory mediators (dysregulated inflammation) is associated with maladaptive lung repair and inability to improve ACM permeability, gas exchange, and lung mechanics over time.

In a phase II randomized controlled trial, Meduri and collaborators tested the hypothesis that prolonged administration of low dose methylprednisolone (1mg/Kg/day) initiated in early severe ARDS (within 72 h of diagnosis) downregulates systemic inflammation and leads to earlier resolution of pulmonary organ dysfunction and a reduction in duration of mechanical ventilation and ICU stay. The pre-defined primary end point to terminate the trial was a 1-point reduction in Lung Injury Score (LIS) or successful extubation by day 7. The duration of treatment was up to 28 days. In intention-to-treat analysis, the response of the two groups (63 treated and 28 control) clearly diverged by day 7 with twice the proportion of treated patients achieving a 1-point reduction in LIS (69.8% vs. 35.7%; P = 0.002) and breathing without assistance (53.9% vs. 25.0%; P = 0.01). Improvement by day 7 correlated with survival by day 7 (R = 0.41; P < 0.001) and hospital survival (R = 0.59; P < 0.001). Treatment was associated with a reduction in the duration of mechanical ventilation (5 vs. 9.5; P = 0.002), ICU stay (7 vs. 14.5; P = 0.007), and ICU mortality (79.4% vs. 57.4%; P = 0.03). At one year, the absolute difference in mortality was 17% (63.5% vs. 46.4%; P = 0.13).

The primary objective of the trial was to test the effect of treatment on lung function; a new larger trial is therefore needed to evaluate the effect of methylprednisolone treatment on survival. The primary aim of the proposed randomized trial is to determine if low-dose methylprednisolone infusion, compared to placebo, will reduce all cause 28-day mortality. Among patients admitted to the ICU with ALI/ARDS, we hypothesize that methylprednisolone infusion will reduce 28-day all cause mortality from 50% to 33% (aggregate data from five randomized studies).

SPECIFICS. In patients with ARDS, the administration of prolonged methylprednisolone treatment will decrease (in comparison to placebo):

* All causes 28-day mortality (primary variable).
* Laboratory indices of systemic inflammation (i.e., C-reactive protein, etc.).
* Physiological and laboratory indices of organ dysfunction.
* Duration of mechanical ventilation and ICU stay. ADDITIONAL SURVIVAL ANALYSIS. - ICU and hospital all cause mortality, defined as the proportion of patients alive in each group at first ICU discharge and hospital discharge.

All patients with ALI/ARDS of less than 72 hrs will be enrolled.

EXIT CRITERIA

1. Development of serious complications attributable to glucocorticoid therapy.

   * Gastrointestinal bleeding requiring transfusion
   * Perforated viscus
   * Fungal infection at more than 2 sites
2. Development of life-threatening conditions (i.e. immune thrombocytopenia, vasculitis, etc.) that necessitate glucocorticoid treatment.

PROTECTION OF RECRUITED SUBJECTS: PREVENTION OF COMPLICATIONS ASSOCIATED WITH GLUCOCORTICOID TREATMENT.In conformity with ethical principles that guide clinical critical care research, the protocol incorporates steps to maximize benefits and to minimize risks (i.e., to secondary prevention of potential complications associated with glucocorticoid treatment) to participants.

A. Treatment-induced blunting of the febrile response. Failed or delayed recognition of nosocomial infections in the presence of a blunted febrile response represents a serious threat to the recovery of patients receiving prolonged glucocorticoid treatment. In conducting a RCT investigating prolonged glucocorticoid treatment, infection surveillance is essential to minimize bias generated by the effect of undiagnosed infections on morbidity/mortality. The study protocol incorporates:

1. Surveillance bronchoscopic or non-bronchoscopic BAL sampling at 5- to 7-day intervals in intubated patients (without contraindication), and
2. Previously described systematic diagnostic protocol if a patient develops:

   * Change in temperature (fever or hypothermia),
   * Increase in immature neutrophil count (≥ 3%)
   * Unexplained increase in minute ventilation (≥ 30%)
   * Unexplained worsening in organ dysfunction (increase in MODS score). The diagnostic protocol includes bronchoscopy, abdominal CT scan, change of central line over wire with cultures of the tip of the catheter, urine and blood cultures. If bilirubin is elevated obtain ultrasound of the gallbladder.

B. Treatment-induced neuromuscular weakness.The combination of prolonged glucocorticoid administration in conjunction with neuromuscular blocking agents may lead to prolonged neuromuscular weakness and delayed weaning. The use of neuromuscular blocking agents is strongly discouraged in this trial.

C. Treatment-induced downregulation of glucocorticoid receptors and rebound inflammation with premature discontinuation of glucocorticoid treatment.Ample experimental and clinical literature support the concept that duration of exposure to glucocorticoids is critical to achieving regulation of cytokine production and demonstrable therapeutic benefits. In experimental ALI, glucocorticoid administration was shown to be effective in decreasing lung collagen and edema formation with prolonged treatment, while premature withdrawal rapidly negated the positive effects of therapy. In patients with unresolving ARDS, premature discontinuation of methylprednisolone administration was associated with physiological deterioration that responded favorably to reinstitution of treatment. Study drug is tapered slowly over time. Since rebound inflammation may occur after termination of treatment, physician use of methylprednisolone is not restricted after completion of treatment with blind study drug.

D. Per os absorption of methylprednisolone is compromised for days after extubation. Yates and collaborators have previously shown undetectable methylprednisolone blood levels when ARDS patients were switched from IV to per os intake of the drug. Although the mechanisms of poor GI absorption following extubation of patients with ARDS are unclear, this factor is clinically relevant and may affect response to treatment. Enteral intake of study drug is postponed to day 5 after extubation.

E. Treatment-induced Hyperglycemia. Hyperglycemia is a known complication of glucocorticoid therapy. An European open randomized clinical trial reported that in surgical patients in the ICU for greater than 5 days, ICU outcome is improved if near-normal glucose control is maintained with insulin therapy. This observation was confirmed in a large observational study of elderly patients admitted to a general ICU. Practice consensus guidelines recommend tight glycemic (< 150 mg/dl) control for septic ICU patients. Glycemia will be monitored every 4-to-6 hours and insulin infusion will be used following recent guidelines- The use of insulin to control glycemia in non-diabetic patients will be recorded .

CONCOMITANT THERAPY. The following concomitant medications are strongly discouraged:

* Neuromuscular blocking agents should be completely avoided,
* Etomidate, especially within the first 24 hours,
* Non-steroidal anti-inflammatory agents.

RANDOMIZATION AND STRATIFICATION. Block randomization stratified according to site is used, and all assignments are made through a central randomization center that generated randomization lists according to the algorithm of Moses-Oakford (RND, Genova, Italy). The randomization ratio will be one active treatment versus one placebo (1:1), with a block size of 3, to receive methylprednisolone infusion or placebo. Patients are prospectively stratified prior to randomization as:

* Intubated versus NPPV treated
* ARDS versus severe ARDS. The purpose of stratification is to distribute equally in both arms intubated versus NPPV treated, and ARDS versus severe ARDS.

ASSIGNMENT OF PATIENTS. A random number generator (a die) will be used to randomize patients. A dynamic allocation scheme is used to stratify patients by

* Initial mode of mechanical ventilation to have an equal distribution in each arm of patients on invasive and noninvasive ventilation,
* Severity of ARDS based on the PaO2:FiO2 response after a 30 min on a standardized ventilator setting with a PEEP of 10.

Study medication will be randomly assigned to numbers in advance. Corticosteroids and placebo will be randomized on a 1:1:1 basis. The random scheme will be prepared in blocks of three. Each patient's eligibility to be entered into the study will be established prior to randomization.

ALLOCATION CONCEALMENT.Only the clinical coordinator is in possession of the sequenced list of treatment assignment for each center. The patients and the investigators are unaware of the patients' treatment assignments. The clinical investigator at each center only assigned a sequential number to each enrolled patient. Assignments for methylprednisolone or placebo infusion are contained in sequentially numbered, opaque, sealed envelopes that are in possession of the recruiting investigator at each center. The recruiting investigator sends the sealed envelopes to the independent pharmacist in charge (or ICU manager) only after the participant's name is written on the appropriately sequenced envelope. The signed sealed envelope are opened and read only by the pharmacists in charge in a separate place.

UNBLINDING. The investigator may unblind the randomization code for a specific patient in case of an emergency and if the proposed therapy to be given to the patient depends on the identification of the treatment given. This possibility is most unlikely and is discouraged, as patients will usually be treated the same way whether the code is broken or not. If the code is broken (by opening a provided sealed envelope), the investigator must communicate via internet or fax a letter within two working days to the Data and Safety Monitoring Committee (DSMC) stating the date, time and reasons for breaking the blinded code. All envelopes will be returned at the end of the study.

SAMPLE SIZE. The sample size depends on the magnitude of the difference in mortality that is considered important. The study is designed to detect an absolute difference in all cause 28-day mortality of 17%, expecting a mortality of 33% and 50% for prolonged methylprednisolone treatment and placebo, respectively. A sample size of at least 400 patients would be required for this clinical trial to detect an improvement data significance level of 0.05 and a power of 0.90, considering an attrition rate of 10%.

ANALYSIS. This study is analyzed as intention-to-treat for patients that receive at least 24 hours of study drug and had no exclusion criteria recognized after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Age. Patients age 18 years or older admitted to the intensive care unit.
* ALI/ARDS criteria. The diagnosis of ALI/ARDS requires all of the following criteria:

  * Respiratory failure requiring mechanical ventilation - via endotracheal intubation or noninvasive positive pressure ventilation
  * Acute onset of bilateral pulmonary densities on chest radiograph in the contest of appropriate predisposing injury or illness with no evidence of left ventricular failure,
  * Static pulmonary compliance < 50 cm H2O
  * Ratio of partial pressure of arterial oxygen to partial pressure of alveolar oxygen (PaO2:FiO2 ) equal or less than 300 (criteria for ALI) or 200 (criteria for ARDS) with FiO2 1.0.
* Severe ARDS. PaO2:FiO2 equal or less than 200 after 30 minutes of standardized ventilatory management on PEEP of 10 cm H2O with FiO2 1.0.

Exclusion Criteria:

* Failure to obtain written informed consent from the patient or a next of kin.
* Trauma-induced ARDS.
* Major gastrointestinal bleeding requiring transfusion of 5 units or more of packed red blood cells (PRBC) within 3 months current hospitalization
* Condition requiring > 0.5mg/Kg/day of prednisone equivalent (i.e., acute asthma or chronic obstructive pulmonary disease [COPD])
* Patients enrolled in another experimental (interventional) protocol within the past 30 days, which might adversely impact on the results of this study as determined by the investigators
* Pregnancy confirmed by urine or serum test
* Weight is > 200% of ideal body weight
* Non-ambulatory resident of long-term care facility
* Primary care physician not committed to full, aggressive support of the patient at the time of randomization
* Moribund patient (i.e., not expected to live more than 24 hr) or with recent (within 7 days or anytime during present hospitalization) cardiopulmonary arrest
* Known or suspected irreversible cessation of all brain function
* Presence of preexisting medical condition which is irreversible and expected to be fatal within 3 months
* Immunosuppression including HIV+ status, history of bone marrow or solid organ transplantation, current malignancy, neutropenia, receiving cytotoxic therapy for any reason, and acute burn injury
* Severe chronic liver disease (Child-Pugh Class C score > 10 points)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-02; Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
The primary aim is to determine if low-dose methylprednisolone infusion, compared to placebo, will reduce all cause 28-day mortality, defined as the proportion of patients alive in each group on study day 28 at midnight. | one year

SECONDARY OUTCOMES:
The secondary aims are the effects of treatment on: a. Systemic inflammation b. Duration of mechanical ventilation c. Multiple organ dysfunction syndrome d. Duration of ICU and hospital stay e. Cardiovascular morbidity-mortality f. Complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Principal Investigator — Catholic University of Sacred Heart, Rome; Umberto Meduri, MD, Study Director — University of Tennessee Health Science Center Memphis, TN, USA
Locations (1):
- UCSC, Policlinico Universitario A. Gemelli, ICU, Rome, Rome, Italy

REFERENCES:
- [Background] Meduri GU, Tolley EA, Chrousos GP, Stentz F. Prolonged methylprednisolone treatment suppresses systemic inflammation in patients with unresolving acute respiratory distress syndrome: evidence for inadequate endogenous glucocorticoid secretion and inflammation-induced immune cell resistance to glucocorticoids. Am J Respir Crit Care Med. 2002 Apr 1;165(7):983-91. doi: 10.1164/ajrccm.165.7.2106014. PMID 11934726
- [Background] Meduri GU, Headley AS, Golden E, Carson SJ, Umberger RA, Kelso T, Tolley EA. Effect of prolonged methylprednisolone therapy in unresolving acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1998 Jul 8;280(2):159-65. doi: 10.1001/jama.280.2.159. PMID 9669790
- [Background] Steinberg KP, Hudson LD, Goodman RB, Hough CL, Lanken PN, Hyzy R, Thompson BT, Ancukiewicz M; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network. Efficacy and safety of corticosteroids for persistent acute respiratory distress syndrome. N Engl J Med. 2006 Apr 20;354(16):1671-84. doi: 10.1056/NEJMoa051693. PMID 16625008
- [Background] Annane D, Sebille V, Bellissant E; Ger-Inf-05 Study Group. Effect of low doses of corticosteroids in septic shock patients with or without early acute respiratory distress syndrome. Crit Care Med. 2006 Jan;34(1):22-30. doi: 10.1097/01.ccm.0000194723.78632.62. PMID 16374152
- [Background] Confalonieri M, Urbino R, Potena A, Piattella M, Parigi P, Puccio G, Della Porta R, Giorgio C, Blasi F, Umberger R, Meduri GU. Hydrocortisone infusion for severe community-acquired pneumonia: a preliminary randomized study. Am J Respir Crit Care Med. 2005 Feb 1;171(3):242-8. doi: 10.1164/rccm.200406-808OC. Epub 2004 Nov 19. PMID 15557131
- [Result] Meduri GU, Golden E, Freire AX, Taylor E, Zaman M, Carson SJ, Gibson M, Umberger R. Methylprednisolone infusion in early severe ARDS: results of a randomized controlled trial. Chest. 2007 Apr;131(4):954-63. doi: 10.1378/chest.06-2100. PMID 17426195